CLINICAL TRIAL: NCT01450228
Title: A Double-blind, Parallel Group, Randomised, Placebo Controlled, Multicenter, Bridging Phase III Study of Efficacy and Safety of KI1001 in the Improvement of Sleep Quality in ≥ 55 Years Old Insomnia Patients
Brief Title: Efficacy and Safety of KI1001 in ≥ 55 Years Old Insomnia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Collaborators: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-CC-8302
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo KI1001 (Placebo Comparator)
  Interventions: Drug: Placebo KI1001
- KI1001 (Experimental)
  Interventions: Drug: KI1001

INTERVENTIONS:
Drug: KI1001 — Prolonged release melatonin 2mg
  Arms: KI1001
Drug: Placebo KI1001 — Placebo KI1001 tablets
  Arms: Placebo KI1001

SUMMARY:
KI1001(Circadin®, Prolonged release tablet which contains melatonin) has showed its efficacy to improve sleep quality in over 55 years old primary insomnia patients. This is a bridging study to investigate the efficacy and safety of KI1001(Circadin®) in Korean patients.

DETAILED DESCRIPTION:
Studies throughout the world have shown that insomnia is a common complaint that occurs in 10-50% of the population depending on age, sex and country. Among the wide variety of available treatments of sleep disturbances, the most commonly prescribed hypnotics are the benzodiazepines (BZD) and non-BZD hypnotics.

However, these hypnotics were often associated with rebound, dependency, tolerance, higher risk of falls mainly in the elderly population, anterograde memory disturbances and increased risk for motor accidents the next day.

In response to the unmet clinical need for a safe and efficacious alternative treatment for primary insomnia, that in addition to treating quantitative sleep problems, would improve sleep quality and daytime functioning, a clinical development program on melatonin for the treatment of primary insomnia was initiated.

This study is conducted using a randomised, double-blind, placebo controlled parallel group design, after a single-blind placebo period. Primary insomnia patients aged over 55 will be screened for entry into the study.

After placebo run-in period, Patients will enter a 3 weeks double-blind treatment period.

Primary parameter is quality of sleep, secondary parameters are including getting to sleep, awakening from sleep, behavior following wakefulness, quality of day and night, sleep latency and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged ≥55 years
* Suffering from primary insomnia according to DSM-IV criteria and for whom this is the consultation complaint
* Good anticipated compliance
* Written informed consent to participate in the study given by the patient voluntarily
* Confirmed diagnosis of primary insomnia by sleep history questionnaire
* Established baseline pathology
* A good compliance during the two-weeks placebo run-in period defined as 70% to 130% of prescribed tablets
* Correct use of the Sleep Diary and of the LSEQ

Exclusion Criteria:

* According to DSM-IV, subjects belonging to the following groups are excluded : 780.59(breathing related sleep disorder); 307.45(circadian thyrhm sleep disorder); 307.47(dyssomnia not otherwise specified); 780.XX(sleep disorder due to a general medical condition)
* Known or suspected hypersensitivity to exogenous melatonin or melatonin receptor agonists
* Known positive serology for human immunodeficiency virus (HIV) I antibodies or HIV II antibodies
* Known chronic active viral hepatitis
* Drug abuse or history or drug abuse(including alcohol)
* History of severe pathology likely to recur during or immediately after the study
* History of severe cardiac disorders
* History of severe neurological disorders or cerebral neurosurgery
* History of severe psychiatric disorders, especially psychosis and depression, sismotherapy
* depression will be assessed by the Raskin scale : a patient with a total score ≥ 6 will not be included
* anxiety will be assessed by the Covi scale : a patient with a total score ≥ 6 will not be included
* dementia will be assessed with the Mini Mental State (MMS) : a patient with a score ≤ 24 or 26 (depending on the socio-educational level of the patient) will not be included
* Neuro-psychiatric pathologies that might interfere with insomnia, patient assessment or study medication
* Use of psychotropic treatments for the past 3 months and during the study
* Use of benzodiazepines or other hypnotics during preceding two weeks (including all benzodiazepines; zopiclone, zolpidem, zaleplon, barbiturates, buspirone and hydroxyzine)
* All hypnotics or treatments used as an hypnotic are not allowed during the study
* Severe pain likely to interfere with sleep
* Other sleep disorders according to DSM-IV criteria identified by numerical ICD 9 code: breathing-related sleep disorder (780.59), circadian rhythm sleep disorder (307.45), dyssomnia not otherwise specified (307.47) and other sleep disorders (780.xx)
* Serious diseases that could interfere with patient assessment
* Organic pathologies which have not stabilised and that might interfere with sleep, patient assessment or study medication
* Intercurrent acute or chronic somatic diseases likely to interact with sleep (for example: chronic pain from any aetiology, benign prostatic hypertrophy likely to require surgery in the coming six months)
* Any concomitant documented progressive disease likely to interfere with the conduct of the study
* Any medical condition which might interfere with the completion of the study, or which would be adversely affected and thereby increasing the risk for the patient or interfering with patient assessments.
* Patients with an excessive consumption of alcohol, coffee or tea
* Patients with an irregular lifestyle or life pattern (e.g. shift workers and patients likely to be jet lagged)
* Patients with a Body Mass Index above 30 - obesity
* Patients who have taken any investigational drug within two months preceding the first dose of the study drug. Investigational drug is defined as any drug for which a marketing authorisation has not been granted in the country where the study was conducted.
* Patients receiving concomitant treatment which are not permitted
* A positive drug screen (benzodiazepines and opiates) during the initial two week placebo run-in period

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
QOS in LSEQ | three weeks
  LSEQ - Leeds Sleep Evaluation Questionnaire QOS - Quality of Sleep

SECONDARY OUTCOMES:
GTS in LSEQ | three weeks
  LSEQ - Leeds Sleep Evaluation Questionnaire GTS - Getting to Sleep
QOD | three weeks
  Quality of day in Patient Diary
WHO 5-welling index | three weeks
PSQI | three weeks
  Pittsburgh Sleep Quality Index
AFS in LSEQ | three weeks
  LSEQ - Leeds Sleep Evaluation Questionnaire AFS - Awakening from Sleep
BFW in LSEQ | three weeks
  LSEQ - Leeds Sleep Evaluation Questionnaire BFW - Behavior following Wakefulness
QON | three weeks
  Quality of Night in Patient Diary

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Sang Yoon, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Jung-Hie Lee, M.D., Ph.D., Principal Investigator — KangWon National University Hospital; Seung-Chul Hong, M.D., Ph.D., Principal Investigator — The Catholic University of Korea, St. Vincent Hospital; Doo-Heum Park, M.D., Ph.D., Principal Investigator — Konkuk University Medical Center; Won-Chul Shin, M.D., Ph.D., Principal Investigator — Kyung Hee University Hospital at Gangdong; In-Young Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Kyu-In Jung, M.D., Ph.D., Principal Investigator — Catholic University of Korea Saint Paul's Hospital; Yong-Won Cho, M.D., Ph.D., Principal Investigator — Keimyung University Dongsan Medical Center; Jee-Hyun Kim, M.D., Ph.D., Principal Investigator — Dankook University; Seock-Hoon Chung, M.D., Ph.D., Principal Investigator — University of Ulsan College of Medicine, Asan Medical Center
Locations (10):
- South Korea (10):
  - Dankook University Hospital, Cheonan, Chungcheongnam
  - Keimyung University, Dongsan Medical Center, Daegu, Daegu
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Chonnam National University Hospital, Gwangju, Gwangju
  - Seoul National University Bundang Hospital, Sungnam, Gyeonggi-do
  - St. Vincent Hospital, Suwon, Gyeonggi-do
  - St. Paul's Hospital, Seoul, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Konkuk University Medical Center, Seoul, Seoul